CLINICAL TRIAL: NCT01932853
Title: Evaluation of the Association of Dialysis Dose Obtained by Kt and Mortality in Hemodialysis Patients
Brief Title: Association Between Dose Dialysis by Kt and Mortality
Status: Completed | Type: Observational
Sponsor: NephroCare Spain (Industry)
Responsible Party: Principal Investigator, Rosa Ramos, MD, Ph, NephroCare Spain
Other Study IDs: QM-RR-02
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2015-10

CONDITIONS: End Stage Renal Disease; Hemodialysis Patients
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis patients: Patients > 18y hemodialysis for at least 6 months at any center of Spain Fresenius Medical Care (FMC) meeting the inclusion criteria.

SUMMARY:
The aim of this study is to assess whether patients receiving current recommendations of an adequate dialysis dose by Kt adjusted for body surface area improved survival at 24 months compared to those who do not get it, as well as assess whether patients receiving a dose greater obtain more benefit.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* > six months on hemodialysis
* Receiving 3 sessions of dialysis per week
* Having 5 or more valid measures of Kt during the month

Exclusion Criteria:

* active chronic inflammatory diseases
* Liver cirrhosis
* Neoplasms
* Chronic immunosuppression or use of anti-inflammatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects:
  Patients> 18 years in hemodialysis treatment at any FMC center of Spain that meet the inclusion criteria.
  Data will be collected according to clinical practice and patients will be categorized according to their dose of Kt, along the two years of the study. Will seek the association of dialysis dose with mortality and hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 6129 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mortality | two years

SECONDARY OUTCOMES:
Hospitalization | two years

OTHER OUTCOMES:
Mortality and hospitalization cause | two years

CONTACTS AND LOCATIONS:
Overall Officials: Francesc Maduell, MD, Ph, Principal Investigator — Servei Nefrologia, ICNU, Hospital Clínic.
Locations (1):
- NephroCare Spain, Madrid, Madrid, Spain